CLINICAL TRIAL: NCT00370955
Title: The Effect of Hydrodynamic Parameters on Corneal Endothelial Cell Loss After Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Ophthalmic Research Center of Shaheed Beheshti Medical University, Shaheed Beheshti Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8527
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2009-12-25 (Estimated); Status verified 2008-10

CONDITIONS: Cataract
Keywords: Phacoemulsification; Corneal endothelial cell loss; Hydrodynamic parameters; Total ultrasound energy; Total infused fluids
MeSH Terms: conditions — Cataract; Corneal Endothelial Cell Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High vacuum group (Active Comparator): Those patients who underwent phacoemulsification using high hydrodynamic parameter: 400 mmHg vacuum and 40 ml/min flow rate.
  Interventions: Procedure: phacoemulsification using either high vacuum or low vacuum techniques
- Low vacuum group (Active Comparator): Patients who underwent phacoemulsification using low hydrodynamic parameters: 200 mmHg vacuum and 20 ml/min flow rate.
  Interventions: Procedure: phacoemulsification using either high vacuum or low vacuum techniques

INTERVENTIONS:
Procedure: phacoemulsification using either high vacuum or low vacuum techniques — All surgeries were performed using Sovereign phacoemulsification system (AMO) using Whitestar technology.
  Other Names: stop and chop technique

SUMMARY:
The purpose of this study is to compare two surgical techniques (high vacuum and low vacuum) on corneal endothelium after phacoemulsification.

DETAILED DESCRIPTION:
Patients aged 50 to 70 years old with moderate lens opacities (nuclear sclerosis of 3+) were included. The exclusion criteria were: 1-previous corneal pathology (dystrophic or degenerative such as Fuchs' endothelial dystrophy or advanced trachoma), 2- pseudoexfoliation syndrome (PEX), 3- history of intra ocular surgery, 4- glaucoma or ocular hypertension, 5- eyes with a history of anterior uveitis, 6- diabetes mellitus, 7- anterior chamber depth (ACD) less than 2.5 mm or more than 4 mm, 8- axial length less than 21 mm or more than 25 mm, 9- density of endothelial cells less than 1500 cells per mm2, 10- polymegatism (CV > 0.4), 11- keratometric astigmatism more than 1.5 Diopters (D), 12- history of contact lens usage, 13- Intra-operative complications (posterior capsule rupture with or without vitreous loss), 14- postoperative uveitis, 15- postoperative surgical wound leakage, 16- deep-set eye, and 17- size of dilated pupil less than 6 mm. Nucleus density was evaluated using the LOCS III classification system Patients were divided in 2 groups randomly: Group 1 included those candidates for phacoemulsification using high hydrodynamic parameter: 400 mmHg vacuum and 40 ml/min flow rate (high vacuum technique) whereas group 2 consisted of patients who underwent phacoemulsification using low hydrodynamic parameters: 200 mmHg vacuum and 20 ml/min flow rate (low vacuum technique). All surgeries were performed by one surgeon using stop and chop technique with sovereign (white star technology) (AMO, USA). During sculpting stage, vacuum was 40mmHg and flow rate is 20ml/min, in both groups. Irrigation aspiration of cortical material and viscoelastic were bimanually and semi automatically performed with flow rate of 30ml/min.

Total ultrasound power and total volume of BSS in both groups were measured. Pachymetry, endothelial cell density, polymegathism, before and 1, 6 and 12 weeks after intervention were also evaluated. Statistically analysis of data included univariate (student t-test and x2) and multivariate (regression model) analysis of postoperative results.

ELIGIBILITY:
Inclusion Criteria were:

* Moderate lens opacity (Nuclear sclerosis 3+)
* Age between 50 to 70 years

The exclusion criteria were:

* Previous corneal pathology (dystrophic or degenerative such as Fuchs' endothelial dystrophy or advanced trachoma),
* Pseudoexfoliation syndrome (PEX),
* History of intra ocular surgery,
* Glaucoma or ocular hypertension,
* Eyes with a history of anterior uveitis,
* Diabetes mellitus,
* Anterior chamber depth (ACD) less than 2.5 mm or more than 4 mm,
* Axial length less than 21 mm or more than 25 mm,
* Density of endothelial cells less than 1500 cells per mm2,
* Polymegatism (CV > 0.4),
* Keratometric astigmatism more than 1.5 Diopters (D),
* History of contact lens usage,
* Intra-operative complications (posterior capsule rupture with or without vitreous loss),
* Postoperative uveitis,
* Postoperative surgical wound leakage,
* Deep-set eye, and 17- size of dilated pupil less than 6 mm.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Total ultrasound energy dissipated to the eye, total infused fluid, Endothelial cell loss | All patients were examined on postoperative day 1 and weeks 1, 6 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Baradaran Raffiee, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Alireza Baradaran Raffiee, Tehran, Tehran Province, Iran

REFERENCES:
- See also: Official webpage of ophthalmic research center of Shahid Beheshti University of Medical Sciences — http://www.orcir.org/english/Default.aspx
- See also: Published article — http://www.ncbi.nlm.nih.gov/pubmed/19304097?itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum&ordinalpos=2